CLINICAL TRIAL: NCT05899738
Title: A Phase 1, Open-Label, Randomized, Two-Part, Two-Period, Two-Sequence Crossover Study to Assess the Relative Bioavailability of Iberdomide (CC-220) Powder for Reconstitution Formulation to the Reference Capsule Formulation and to Assess the Effect of Food on the Pharmacokinetics of Powder for Reconstitution Formulation in Healthy Adult Participants
Brief Title: A Study to Compare the Relative Bioavailability of Two Iberdomide (CC-220) Formulations and to Assess The Effect Of Food on the Drug Levels of Iberdomide in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM048-1038
Record Dates: First submitted 2023-05-17; First posted 2023-06-12 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteers
Keywords: Healthy; Iberdomide; Bioavailability; Crossover; Powder Formulation; Food Effect; Fed; Fasted
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — iberdomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Iberdomide Powder (Fasted), followed by Iberdomide Capsule (Fasted) (Experimental)
  Interventions: Drug: Iberdomide
- Iberdomide Capsule (Fasted), followed by Iberdomide Powder (Fasted) (Experimental)
  Interventions: Drug: Iberdomide
- Iberdomide Powder (Fasted), followed by Iberdomide Powder (Fed) (Experimental)
  Interventions: Drug: Iberdomide
- Iberdomide Powder (Fed), followed by Iberdomide Powder (Fasted) (Experimental)
  Interventions: Drug: Iberdomide

INTERVENTIONS:
Drug: Iberdomide — Specified dose on specified days
  Other Names: BMS-986382; CC-220

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability for the new iberdomide powder for reconstitution formulation relative to the reference capsule formulation and to assess the effect of food on the pharmacokinetics of powder for reconstitution formulation in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 18.0 to 33.0 kilograms (kg)/square meter, inclusive, and body weight ≥50 kg.
* A female participant is eligible to participate if she is not of childbearing potential as defined in the protocol.
* Males who are sexually active with woman of childbearing potential must agree to follow instructions for method(s) of contraception as described in the protocol and included in the informed consent form.
* Male participants are required to use a condom and must refrain from donating sperm during the intervention period and for at least 28 days after the last dose of study intervention.

Exclusion Criteria:

* Any significant acute or chronic medical illness.
* Current or recent (within 3 months of the first dose of the investigational medicinal product) gastrointestinal disease or procedure that could possibly affect drug absorption, distribution, metabolism, and excretion (for example, bariatric procedure).
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, electrocardiogram, or clinical laboratory determinations.
* Female who are of childbearing potential and females who are breastfeeding.

Note: Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to 72 hours post-dose for Period 1 and Period 2 (each period is 4 days, with a 5-9 day washout between each dose)
Area Under the Plasma Concentration-time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUC(0-T)) | Up to 72 hours post-dose for Period 1 and Period 2 (each period is 4 days, with a 5-9 day washout between each dose)
Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinite Time (AUC(INF)) | Up to 72 hours post-dose for Period 1 and Period 2 (each period is 4 days, with a 5-9 day washout between each dose)

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Up to 28 days
Number of Participants with Vital Sign Abnormalities | Up to 20 days
Number of Participants with Clinical Laboratory Abnormalities | Up to 20 days
Number of Participants with Electrocardiogram Abnormalities | Up to 20 days
Number of Participants with Physical Examination Abnormalities | Up to 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT05899738.html